CLINICAL TRIAL: NCT07117981
Title: Treatment of Graves' Orbitopathy in Patients Failing Corticosteroid Therapy: Multicenter National Retrospective Study- Basedow
Brief Title: Describe the Progression of Inflammatory Orbitopathy and the Biological Progression of Patients Receiving Second-line Treatment
Acronym: HZN-IIT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Other Study IDs: P23-05
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Basedow Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Describe the progression of inflammatory orbitopathy and the biological progression of patients receiving second-line treatment (immunosuppressants, radiotherapy, or biotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older with moderate to severe orbitopathy;
* Patients followed in endocrinology with the goal of achieving euthyroidism;
* Corticosteroid-resistant patients: patients who have received at least 3 weeks of treatment with 500 mg weekly corticosteroid boluses and have not shown improvement in the clinical activity score (CAS);
* Corticosteroid-dependent patients: relapse with a CAS of 3 or higher when decreasing or stopping corticosteroid therapy;
* Patients with a CAS ≥ 3 or CAS <3 with moderate to severe orbitopathy (according to EUGOGO);
* Patients treated with immunotherapy, biotherapy, or radiotherapy as second-line treatment;
* Patients who are not opposed to the reuse of their health data.

Exclusion Criteria:

* Patients who have undergone bone or fat decompression surgery;
* Patients with severe corneal involvement (Grade B or C; NO SPECS classification);
* Patients with optic neuropathy (Grade B and C; NO SPECS classification);
* Patients who have received 1 gram corticosteroid boluses for dysthyroid orbitopathy;
* Patients who have opposed the reuse of their health data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data collection concerns patients with Graves' orbitopathy who have received corticosteroid treatment and second-line treatment (immunosuppressants, biotherapy) since 2015, 2021, or 2022. A decision was made to limit the inclusion to patients who started second-line treatment between January 2022 and December 2023, with clinical follow-up until the end of 2024, in order to limit selection bias and ensure an adequate follow-up period.
  The inclusion period extends until June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Response to second-line basedow treatment | Patients who started a second-line treatment between January 2022 and December 2023, with clinical follow-up until the end of 2024, were included in order to minimize selection bias. inclusion period: until december 2025
  Practices in France regarding the use of these second-line treatments appear to be heterogeneous, and their effectiveness has never been compared through randomized studies.
  investigators propose to collect and analyze the therapeutic outcomes of second-line treatment in patients with Graves' orbitopathy. The data collection concerns patients with Graves' orbitopathy who have received corticosteroid therapy and a second-line treatment (immunosuppressant, biotherapy) since 2022.
  Data from the medical records of patients included.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, paris
  - CHU Caen Normandie COTE DE NACRE, Caen
  - CHU Lyon - Hospices Civils de Lyon, Lyon
  - Hopital Saint Joseph, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Nîmes, Nîmes
  - Hopital Fondation de Rothschild, Paris
  - CHU de Pontchaillou, Rennes
  - Hopital Civil / Nouvel Hopital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No
Each center remains the owner of its data, so it is possible to extract and send data from each center via the eCRF for theses or publications

REFERENCES:
- [Background] Chin YH, Ng CH, Lee MH, Koh JWH, Kiew J, Yang SP, Sundar G, Khoo CM. Prevalence of thyroid eye disease in Graves' disease: A meta-analysis and systematic review. Clin Endocrinol (Oxf). 2020 Oct;93(4):363-374. doi: 10.1111/cen.14296. Epub 2020 Aug 10. PMID 32691849
- [Background] Bartalena L, Baldeschi L, Dickinson A, Eckstein A, Kendall-Taylor P, Marcocci C, Mourits M, Perros P, Boboridis K, Boschi A, Curro N, Daumerie C, Kahaly GJ, Krassas GE, Lane CM, Lazarus JH, Marino M, Nardi M, Neoh C, Orgiazzi J, Pearce S, Pinchera A, Pitz S, Salvi M, Sivelli P, Stahl M, von Arx G, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). Consensus statement of the European Group on Graves' orbitopathy (EUGOGO) on management of GO. Eur J Endocrinol. 2008 Mar;158(3):273-85. doi: 10.1530/EJE-07-0666. No abstract available. PMID 18299459
- [Background] Bartalena L, Kahaly GJ, Baldeschi L, Dayan CM, Eckstein A, Marcocci C, Marino M, Vaidya B, Wiersinga WM; EUGOGO dagger. The 2021 European Group on Graves' orbitopathy (EUGOGO) clinical practice guidelines for the medical management of Graves' orbitopathy. Eur J Endocrinol. 2021 Aug 27;185(4):G43-G67. doi: 10.1530/EJE-21-0479. PMID 34297684
- [Background] Vargas-Uricoechea H. Autoimmune Thyroid Disease and Differentiated Thyroid Carcinoma: A Review of the Mechanisms That Explain an Intriguing and Exciting Relationship. World J Oncol. 2024 Feb;15(1):14-27. doi: 10.14740/wjon1728. Epub 2023 Dec 9. PMID 38274715
- [Background] Lee JY, Lee MK, Lee JH, Kim K, Bae K, Sohn SY. Cancer Risks of Patients with Graves' Disease Who Received Antithyroid Drugs as Initial Treatment: A Nationwide Population-Based Analysis. Thyroid. 2024 Oct;34(10):1271-1279. doi: 10.1089/thy.2024.0178. Epub 2024 Sep 23. PMID 39228052
- [Background] Goodman RS, Johnson DB, Balko JM. Corticosteroids and Cancer Immunotherapy. Clin Cancer Res. 2023 Jul 14;29(14):2580-2587. doi: 10.1158/1078-0432.CCR-22-3181. PMID 36648402
- [Background] Prummel MF, Bakker A, Wiersinga WM, Baldeschi L, Mourits MP, Kendall-Taylor P, Perros P, Neoh C, Dickinson AJ, Lazarus JH, Lane CM, Heufelder AE, Kahaly GJ, Pitz S, Orgiazzi J, Hullo A, Pinchera A, Marcocci C, Sartini MS, Rocchi R, Nardi M, Krassas GE, Halkias A. Multi-center study on the characteristics and treatment strategies of patients with Graves' orbitopathy: the first European Group on Graves' Orbitopathy experience. Eur J Endocrinol. 2003 May;148(5):491-5. doi: 10.1530/eje.0.1480491. PMID 12720530